CLINICAL TRIAL: NCT02891603
Title: A Phase I/II GVHD Prevention Trial Combining Pacritinib With Sirolimus-Based Immune Suppression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: CTI BioPharma (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18783; 5R01HL133823-02 (NIH)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Graft Vs Host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Tyrosine Kinase Inhibitors; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1, Level 1: Pacritinib with Sirolimus and Tacrolimus (Experimental): After standard of care allogenic hematopoietic cell transplantation, Pacritinib will be added to standard treatment with Sirolimus and Tacrolimus (PAC/SIR/TAC).
  100 mg Pacritinib will begin taken by mouth the day of the participant's transplant (Day 0) and will continue until 70 days after the transplant..
  Sirolimus will be given the day before transplant and continued daily for at least one year.
  Tacrolimus will begin 3 days before transplant and will be given for at least 50 days.
  Interventions: Drug: Pacritinib; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Allogenic hematopoietic cell transplant (alloHCT)
- Phase 1, Level 2: Pacritinib with Sirolimus and Tacrolimus (Experimental): After standard of care allogenic hematopoietic cell transplantation, Pacritinib will be added to standard treatment with Sirolimus and Tacrolimus (PAC/SIR/TAC).
  100 mg Pacritinib will begin taken by mouth twice daily starting the day of the participant's transplant (Day 0) and continuing until 70 days after the transplant..
  Sirolimus will be given the day before transplant and continued daily for at least one year.
  Tacrolimus will begin 3 days before transplant and will be given for at least 50 days.
  Interventions: Drug: Pacritinib; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Allogenic hematopoietic cell transplant (alloHCT)
- Phase 2: Pacritinib with Sirolimus and Tacrolimus (Experimental): After standard of care allogenic hematopoietic cell transplantation, Pacritinib will be added to standard treatment with Sirolimus and Tacrolimus (PAC/SIR/TAC).
  Patients will take Pacritinib at the MTD: 100 mg Pacritinib will begin taken by mouth twice daily starting the day of the participant's transplant (Day 0) and continuing until 70 days after the transplant..
  Sirolimus will be given the day before transplant and continued daily for at least one year.
  Tacrolimus will begin 3 days before transplant and will be given for at least 50 days.
  Interventions: Drug: Pacritinib; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Allogenic hematopoietic cell transplant (alloHCT)

INTERVENTIONS:
Drug: Pacritinib — Pacritinib Dose and Schedule: 200 mg twice a day (BID) orally from day 0 until day +100. PAC will be tapered to 50% of the total dose at day +70, then 25% of total dose at day +84, then stop at day +100 (+/- 7 days).
  Other Names: PAC; tyrosine kinase inhibitor (TKI)
Drug: Sirolimus — Sirolimus (SIR) will be administered and dosed according to Moffitt Cancer Center, Department of Blood and Marrow Transplantation standard practice. Attending physician discretion is permitted with regard to timing, rapidity, and completion of SIR taper. SIR levels will be monitored according to program standard operating procedures. Dose modifications of SIR for concurrent use of CYP3A4 inhibitors or inducers will be based on program standard operating procedures.
  Other Names: Rapamune
Drug: Tacrolimus — Tacrolimus (TAC) will be administered and dosed according to Moffitt Cancer Center, Department of Blood and Marrow Transplantation standard practice. Attending physician discretion is permitted with regard to timing, rapidity, and completion of TAC taper. TAC levels will be monitored according to program standard operating procedures. Dose modifications of TAC for concurrent use of CYP3A4 inhibitors or inducers will be based on program standard operating procedures.
  Other Names: Prograf
Procedure: Allogenic hematopoietic cell transplant (alloHCT) — Patients will undergo allogenic hematopoietic cell transplant (alloHCT) as a part of their standard of care treatment.

SUMMARY:
The purpose of this study is to examine a new approach to preventing a serious problem after transplant called graft vs. host disease (abbreviated as GVHD).

This is a 3 arm sequential phase I/II, study of Pacritinib with Sirolimus and Tacrolimus (PAC/SIR/TAC) for the prevention of acute GVHD after matched related and unrelated allogeneic hematopoietic cell transplantation (alloHCT).

DETAILED DESCRIPTION:
GVHD is a common problem that occurs after transplant despite the use of standard immune suppressive medications (these are called sirolimus and tacrolimus). GVHD can result in skin rash, nausea, vomiting, diarrhea, and liver damage. Severe GVHD can be life-threatening.

In this study, investigators will add a medication called pacritinib to the combination of sirolimus and tacrolimus to see if this approach can more effectively prevent GVHD. Pacritinib is a medicine used to treat a disease of the bone marrow called myelofibrosis Pacritinib turns off a switch in cells called Janus Kinase 2 (JAK2). Pacritinib is an investigational medicine used in several clinical trials and not FDA approved. JAK2 is an important regulator of inflammation. This inflammation is thought to contribute to GVHD. Pacritinib is able to turn this inflammation off by inhibiting JAK2. Research has shown that blocking JAK2 prevents GVHD in mice and also reduces severe GVHD in transplant patients. Doctors at Moffitt have identified that inflammation from JAK2 is an important cause of GVHD, and is present well before patients develop GVHD symptoms. This trial will study how well pacritinib turns off inflammation during the transplant and if it prevents GVHD when added to our standard medicines.

Pacritinib will begin the day of the participant's transplant (Day 0) and will continue until 70 days after the transplant.

Sirolimus will be given the day before transplant and continued daily for at least one year.

Tacrolimus will begin 3 days before transplant and will be given for at least 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have an available 8/8 HLA-A, -B, -C, and -DRB1 matched-related or unrelated donor allogeneic hematopoietic peripheral blood stem cell graft.
* Signed informed consent.
* Acute myeloid leukemia, myelodysplasia, acute lymphoblastic leukemia, chronic myeloid leukemia, chronic lymphocytic leukemia, myeloproliferative neoplasms, Hodgkin lymphoma, or non-Hodgkin lymphoma requiring a matched allogeneic hematopoietic stem cell transplantation (HSCT). Acute Leukemia (AML or ALL) must be in complete remission defined as: <5% marrow blasts with no morphologic evidence of leukemia, no peripheral blasts, marrow >20% cellular, and peripheral absolute neutrophil count >1000/uL (platelet recovery is not required). Myelodysplasia (MDS) and chronic myeloid leukemia (CML): Must have <5% marrow blasts. Myeloproliferative neoplasms (MPN): Must have <5% peripheral / marrow blasts. Note: Prior use of a JAK2 inhibitor is allowed up to 4 weeks before day 0 of alloHCT. Hodgkin and non-Hodgkin lymphoma: Must have chemosensitive disease.
* Adequate vital organ function.
* Performance status: Karnofsky Performance Status Score ≥ 80%.

Donor Eligibility:

* Eligible donors will include healthy sibling, relative or unrelated donors that are matched with the patient at HLA-A, B, C, and DRB1 by high resolution typing as defined by the Collaborative Trials Network.

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy.
* History of HIV, hepatitis B, or active hepatitis C infection.
* Anti-thymocyte globulin, alemtuzumab, bortezomib, or post-transplant cyclophosphamide as part of GVHD prophylaxis.
* Sorror's co-morbidity factors with total score >4.
* Any patient anticipating or scheduled to receive a tyrosine kinase inhibitor, FLT3 inhibitor, or JAK2 inhibitor (outside of this study) post-HCT.
* QTc>450ms per Fridericia's correction.
* Thrombin time (TT), prothrombin time (PT), or partial thromboplastin time (PTT) >2x upper limit of normal (ULN).
* Grade 3 or higher recent (within the past 6 months) or ongoing non-QTc cardiac adverse events/comorbidities.
* Grade 3 or higher recent or ongoing cardiac dysrhythmias, family history of long QT.

syndrome, or serum potassium <3.0 mEq/L that is persistent and refractory to correction.

* Grade 3 or higher recent or ongoing bleeding events.
* Symptomatic or uncontrolled cardiovascular disease, myocardial infarction or severe/unstable angina within the past 6 months, or New York Heart Association (NYHA) Class III or IV congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pidala, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Pidala J, Walton K, Elmariah H, Kim J, Mishra A, Bejanyan N, Nishihori T, Khimani F, Perez L, Faramand RG, Davila ML, Nieder ML, Sagatys EM, Holtan SG, Lawrence NJ, Lawrence HR, Blazar BR, Anasetti C, Sebti SM, Betts BC. Pacritinib Combined with Sirolimus and Low-Dose Tacrolimus for GVHD Prevention after Allogeneic Hematopoietic Cell Transplantation: Preclinical and Phase I Trial Results. Clin Cancer Res. 2021 May 15;27(10):2712-2722. doi: 10.1158/1078-0432.CCR-20-4725. Epub 2021 Mar 22. PMID 33753457
- [Derived] Betts BC, Bastian D, Iamsawat S, Nguyen H, Heinrichs JL, Wu Y, Daenthanasanmak A, Veerapathran A, O'Mahony A, Walton K, Reff J, Horna P, Sagatys EM, Lee MC, Singer J, Chang YJ, Liu C, Pidala J, Anasetti C, Yu XZ. Targeting JAK2 reduces GVHD and xenograft rejection through regulation of T cell differentiation. Proc Natl Acad Sci U S A. 2018 Feb 13;115(7):1582-1587. doi: 10.1073/pnas.1712452115. Epub 2018 Jan 30. PMID 29382747
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1, Level 1: Pacritinib With Sirolimus and Tacrolimus | Phase 1, Level 2: Pacritinib With Sirolimus and Tacrolimus | Phase 2: Pacritinib With Sirolimus and Tacrolimus
Started | 10 | 8 | 22
Completed | 10 | 8 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Level 1: Pacritinib With Sirolimus and Tacrolimus | Phase 1, Level 2: Pacritinib With Sirolimus and Tacrolimus | Phase 2: Pacritinib With Sirolimus and Tacrolimus | Total
Number analyzed (Participants) | 10 | 8 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 10 | 22
  >=65 years | 2 | 4 | 12 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 9 | 17
  Male | 5 | 5 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 9 | 7 | 21 | 37
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 8 | 22 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: STAT Activity
Description: STAT3 activity in circulating CD4+ T-cells. This is equivalent to 5.5 tablespoons of blood for each assessment. Peripheral blood mononuclear cells (PBMC) will be isolated by Ficoll density gradient. PBMCs will be stimulated with IL-6 for 20 minutes to activate STAT3. Phosphoproteins will be analyzed within T-cells by flow cytometry.
  Result reported is %pSTAT3+CD4+T cells at day +21.
Time Frame: up to 21 days
Population: Evaluable participants treated at MTD (Phase 1 level 2 & Phase 2). Phase 1 level 1 participants were not analyzed for efficacy, therefore there were not included in the analysis population.
Measure: Mean (Standard Deviation); unit: %pSTAT3+CD4+T cells at day +21
Groups:
- Pacritinib With Sirolimus and Tacrolimus: Patients treated with Pacritinib combined with Sirolimus and Tacolimus at Phase 1 Level 2 dose/Phase 2 dose (MTD)
Arm/Group | Pacritinib With Sirolimus and Tacrolimus
Number analyzed (Participants) | 28
%pSTAT3+CD4+T cells at day +21 | 9.623 (10.01)

2. Secondary Outcome: Incidence of Acute GVHD
Description: Cumulative incidence of acute GVHD . Participants will be monitored for clinical signs of acute GVHD. Acute GVHD will be graded per the 1995 consensus guidelines.
Time Frame: up to 100 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pacritinib With Sirolimus and Tacrolimus at MTD: Patients treated with Pacritinib combined with Sirolimus and Tacolimus at Phase 1 Level 2 dose/Phase 2 dose (MTD)
Arm/Group | Pacritinib With Sirolimus and Tacrolimus at MTD
Number analyzed (Participants) | 28
percentage of participants | 46.4 [27.1 to 63.7]

ADVERSE EVENTS:
Time Frame: Adverse events collected from first dose of study drug until 30 days after continuation of study drug, an average of 105 days.
Arm/Group | Phase 1, Level 1: Pacritinib With Sirolimus and Tacrolimus | Phase 1, Level 2: Pacritinib With Sirolimus and Tacrolimus | Phase 2: Pacritinib With Sirolimus and Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/8 | 5/22
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/8 | 8/22
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Level 1: Pacritinib With Sirolimus and Tacrolimus (N=10) | Phase 1, Level 2: Pacritinib With Sirolimus and Tacrolimus (N=8) | Phase 2: Pacritinib With Sirolimus and Tacrolimus (N=22)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
LVEF decrease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Increase in cardiac enzymes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Colitis -Clostridium difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — VOD
Alanine aminotransferase increased - VOD (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased - suspected VOD (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection -Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Erythroderma -acute GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Myocardial infarction as a result of severe acute GVHD
Mulit-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute GVHD of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache -migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Metabolism and Nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Failure to thrive secondary to lack of caregiver support
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Bowel distension and pneumatosis, suspected ischemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Level 1: Pacritinib With Sirolimus and Tacrolimus (N=10) | Phase 1, Level 2: Pacritinib With Sirolimus and Tacrolimus (N=8) | Phase 2: Pacritinib With Sirolimus and Tacrolimus (N=22)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 5 | 5 (12)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 0 (0) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
C Diff (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Suspected VOD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 8 (10) | 10 (14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (4)
Platelet count decreased (Investigations) | 2 (3) | 1 (3) | 8 (11)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (1) | 5 (8)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (14)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
LDH Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CMV+ (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 1 (2)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 5 (5) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 4 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5) | 5 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Folicular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Diffuse rash on face, trunk, and extremities; eyelids swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash over body (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin sloughing off (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 5 (5) | 4 (5)
Edema face (General disorders) | 0 (0) | 2 (3) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel distension and pneumotosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (5) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral fungus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Strep oralis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
C Diff (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Encephalitis - HHV6 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremors (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
BNP High (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02891603/Prot_SAP_000.pdf